CLINICAL TRIAL: NCT00538798
Title: PET Imaging of Brain mGluR5 Receptors Using [18F]SP203 and [11C]SP203
Brief Title: PET Imaging of Brain mGluR5 Receptors Using [18F]SP203
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 070082; 07-M-0082
Record Dates: First submitted 2007-10-02; First posted 2007-10-03 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2015-03-17

CONDITIONS: Healthy; Glutamate Receptor; mGlur5 Protein; Excitatory Amino Acid Receptors; Drug Kinetics; PET Scan
Keywords: Pharmacokinetics; Binding Potential; Glutamate; Positron Emission Tomography; Metabolic Glutamate Receptors; Healthy Volunteer; HV

INTERVENTIONS:
Drug: [18F]SP203

SUMMARY:
The metabotropic glutamate subtype five (mGluR5) receptor is a protein found in the brain and is the target for the excitatory chemical messenger glutimate. The purpose of this protocol is to measure mGluR5 receptors in the brain using positron emission tomography (PET) and a research drug called [18F]SP203.

DETAILED DESCRIPTION:
Metabotropic glutamate receptors are G-protein coupled receptors that respond to glutamate by activating proteins inside nerve cells that affect cell metabolism, thereby fine-tuning the signals sent between cells to maintain balance in neuronal activity. Metabotropic Glutamate receptors (mGluR5) are Group I receptors localized post-synaptically and found in several regions of the brain including the striatum, hippocampus, amygdala, and cortex. Activation of mGluR5 stimulates phospholipase C, resulting in phosphoinositide hydrolysis and increase of intracellular Ca2+ levels. Several potent antagonists for mGluR5 have been developed, including 6 methyl-2-(phenylethynyl)pyridine (MPEP) and 3-[(2-methyl-1,3-thiazol-4yl)ethynyl] pyridine (MTEP) however, no simple derivatives of MPEP or MTEP had proven to be useful for in vivo imaging.

In the present protocol, we will use a new PET ligand [(18)F]SP203 for two reasons: Part 1.) we will perform kinetic brain imaging to quantify mGluR5 binding parameters in brain and determine the reliability and reproducibility of these measures in 15 healthy controls Part 2.) if the tracer is proved successful in the part 1, we plan to estimate radiation-absorbed doses of [(18)F]SP203 in healthy human subjects by performing whole body imaging.

We will also use another new ligand, [11C]SP203, which has the same structure as [(18)F]SP203 but labeled with (11)C instead of (18)F. Part 3) the same purpose as part 1 but with [(11)C]SP203 instead of [(18)F]SP203. Part 4) if [(11)C]SP203 is proved successful in the part 3, we plan to estimate radiation absorbed doses of [(11)C]SP203 in healthy human subjects. At this moment, we do not plan to perform additional scans of [(18)F]SP203 under the current protocol. All future subjects will participate in scans of [(11)C]SP203.

Additionally, Part 5) we will measure the difference in [(18)F]SP203 concentration between the artery and the vein without PET scanning to assess whether the venous blood is a valid and less invasive substitute of arterial blood. In some of [(18)F]SP203 scans performed in the current protocol, we compared [(18)F]SP203 levels between radial artery and antecubital vein and observed 30% - 60% lower levels in vein. We plan to test whether sampling from a vein in the hand and / or warming up makes [(18)F]SP203 levels in vein similar to artery.

Successful development of a PET ligand to image mGluR5 will have a strong impact on clinical management of brain disorders with disruptions in glutamatergic transmission such as schizophrenia, anxiety, and neurodegenerative disorders including Alzheimer s and Parkinson s disease.

ELIGIBILITY:
* INCLUSION CRITERIA:

Healthy control subjects aged 18 65 years, with history/physical exam, ECG, and laboratory tests within one year of the PET scan within normal limits.

EXCLUSION CRITERIA:

1. Current psychiatric illness, substance abuse or severe systemic disease based on history and physical exam.
2. Laboratory tests with clinically significant abnormalities.
3. Prior participation in other research protocols or clinical care in the last year such that radiation exposure would exceed the annual limits.
4. Pregnancy and breast feeding.
5. Claustrophobia. (part 1 and 3 only)
6. Presence of ferromagnetic metal in the body or heart pacemaker. (part 1 and 3 only)
7. Positive HIV test.
8. Consumed alcohol within 48 hours before the PET scan.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-09-28; Study Completion 2015-03-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Masahiro Fujita, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Brodkin J, Bradbury M, Busse C, Warren N, Bristow LJ, Varney MA. Reduced stress-induced hyperthermia in mGluR5 knockout mice. Eur J Neurosci. 2002 Dec;16(11):2241-4. doi: 10.1046/j.1460-9568.2002.02294.x. PMID 12473093
- [Background] Cosford ND, Roppe J, Tehrani L, Schweiger EJ, Seiders TJ, Chaudary A, Rao S, Varney MA. [3H]-methoxymethyl-MTEP and [3H]-methoxy-PEPy: potent and selective radioligands for the metabotropic glutamate subtype 5 (mGlu5) receptor. Bioorg Med Chem Lett. 2003 Feb 10;13(3):351-4. doi: 10.1016/s0960-894x(02)00997-6. PMID 12565928
- [Background] Fujita M, Seibyl JP, Verhoeff NP, Ichise M, Baldwin RM, Zoghbi SS, Burger C, Staley JK, Rajeevan N, Charney DS, Innis RB. Kinetic and equilibrium analyses of [(123)I]epidepride binding to striatal and extrastriatal dopamine D(2) receptors. Synapse. 1999 Dec 15;34(4):290-304. doi: 10.1002/(SICI)1098-2396(19991215)34:43.0.CO;2-B. PMID 10529723